CLINICAL TRIAL: NCT04341623
Title: Epidermal Permeability Barrier Function and Stratum Corneum Hydration of Xerosis Following Application of a Topical Moisturizer
Brief Title: Xerosis and Use of Topical Moisturizer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: IRB00062695
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Xerosis Due to Atopic Dermatitis

STUDY DESIGN:
Intervention Model Description: All three arms will be done at one time
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Other): All patients will receive Cetaphil Pro Eczema moisturizer equipped with an electronic monitor to measure adherence to daily treatment of xerosis
  Interventions: Other: Cetaphil Pro Eczema moisturizer
- Digital Interaction Group (Other): The digital interaction group will receive a survey by email each week asking about their Cetaphil use in addition to the electronic monitor measuring the adherence.
  Interventions: Other: Cetaphil Pro Eczema moisturizer; Behavioral: Electronic interaction
- GPSkin group (Other): The patients in the GPSkin group will receive the GPSkin Barrier® to measure the moisture level of their inner wrist, inner elbow, and dorsal hand daily.
  Interventions: Other: Cetaphil Pro Eczema moisturizer; Behavioral: GPSkin

INTERVENTIONS:
Other: Cetaphil Pro Eczema moisturizer — All 30 patients to receive
Behavioral: Electronic interaction — 10 patients to electronic surveys about moisturizer use
  Arms: Digital Interaction Group
Behavioral: GPSkin — Measuring moisture in the skin
  Arms: GPSkin group

SUMMARY:
The primary hypothesis is that routine measurement of trans epidermal water loss (TEWL) rates and stratum corneum (SC) hydration levels will promote patient adherence to maintenance moisturizer therapy and prevent disease relapse. The project will consist of a trial in which thirty subjects with xerosis receive moisturizer therapy and are randomized to receive either no intervention, a weekly electronic survey to assess patient's response to daily moisturizer, or daily monitoring of the effectiveness of a moisturizer with a portable hydration measurement device. The study team will measure adherence to daily moisturizer use objectively in all three groups with electronic monitors attached to the containers of the moisturizer. The adherence measure will allow the study determine how well moisturizers work for xerosis when that are well used. The study team anticipate that in the no intervention group, adherence will be abysmal and that in the group reporting their response to treatment weekly, adherence will be much better. This will give the study team negative and positive controls for assessing the effect of home barrier monitoring on treatment adherence.

DETAILED DESCRIPTION:
Adult subjects will be offered an opportunity to participate in the study. Subjects will have a diagnosis of xerosis in the context (current or historic) of atopic dermatitis. A total of 30 subjects will be enrolled. After consent and basic demographics, a study team member will use the GPSkin Barrier® device to measure the baseline moisture level of the inner wrist, inner elbow, and dorsal hand of all subjects. Subjects will also fill out questionnaires pertaining to quality of life, measures of predictors of adherence, and severity of xerosis.

Subjects will be randomized into one of three arms: the control group (n= 10), the electronic interaction group to assess patient's response to daily moisturizer (n=10), or the GPSkin group (n=10). All patients will receive Cetaphil Pro Eczema moisturizer equipped with an electronic monitor to measure adherence to daily treatment of xerosis. The digital interaction group will receive a survey by email each week asking about their Cetaphil use. The patients in the GPSkin group will receive the GPSkin Barrier® to measure the moisture level of their inner wrist, inner elbow, and dorsal hand daily. Subjects will be instructed to use the Cetaphil once daily. Subjects will return at 3 months. At this visit, the data from the electronic adherence monitoring will be downloaded, the Cetaphil will be weighed, the patient will fill out the same questionnaires (quality of life, measures of predictors of adherence, and severity of xerosis), and the stratum corneum hydration level will be measured. The intervention subjects will be evaluated on their use of the GPSkin Barrier® to measure their stratum corneum hydration

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older.
* Subject has a working knowledge of English.
* Subject with a diagnosis of xerosis in the context (current or historic) of atopic dermatitis

Exclusion Criteria:

* Subjects under 18 years of age.
* Subject does not have a working knowledge of English.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Xerosis Severity | At Baseline
  Dry Skin/Ichthyosis Area and Severity Index (DASI)
Xerosis Severity | Change from Baseline to 3 months
  Dry Skin/Ichthyosis Area and Severity Index (DASI)
Adherence - Moisturizer | 3 months
  MEMs data of daily use of moisturizer
Adherence - Moisturizer | Baseline
  Weight of moisturizer
Adherence - Moisturizer | Change from baseline to 3 months
  Weight of moisturizer
Transepidermal water loss (TEWL) rates | Baseline
  Use of the GPSkin Barrier device a portable hydration measurement device that measures TEWL rates
Transepidermal water loss (TEWL) rates | Change from baseline to 3 month
  Use of the GPSkin Barrier device a portable hydration measurement device that measures TEWL rates

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Department of Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
Team will determine what will be shared at later time